CLINICAL TRIAL: NCT01093625
Title: Assessment of Daily Disposable Silicone Hydrogel Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0916
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Narafilcon B Contact Lens (Experimental): Investigational Silicone Hydrogel Contact Lens
  Interventions: Device: Narafilcon B Contact Lens
- Spectacles (Active Comparator)
  Interventions: Device: Spectacles

INTERVENTIONS:
Device: Narafilcon B Contact Lens
  Other Names: Investigational Silicone Hydrogel
  Arms: Narafilcon B Contact Lens
Device: Spectacles — spectacle wearers
  Arms: Spectacles

SUMMARY:
The purpose of this study is to evaluate the effect of an investigational silicone hydrogel soft contact lens on new contact lens wearers (neophytes) compared to a control of spectacle wearers.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, comprehend and sign an informed consent (or parental consent/subject assent, as appropriate).
* Willing to comply with the study visit schedule.
* Ages 15 to 39.
* Has access to a cellular telephone with text messaging capabilities.
* Has a current pair of spectacles.
* 'Neophyte' - In this work, 'neophyte' will be taken to mean any subject who has never been dispensed contact lenses. A subject who has taken part in a non-dispensing clinical study or has been fitted with contact lenses in practice but never went on to actually wear the lenses, will also be classified as a 'neophyte'.
* Spherical contact lens (CL) prescription between -0.75D and -6.00D and spectacle cylinder equal to or less than 0.75 DC.
* Monocular best-corrected distance visual acuity (VA) ≥ 20/30 Snellen in each eye.
* Subject agrees to "intent" of wearing the CLs at minimum 6 hours/day for at least 4 days per week.
* They agree not to participate in other clinical research during the duration of this study.

Exclusion Criteria:

* Active ocular allergy, infection, injury, inflammation, or abnormality (e.g., keratoconus) that might interfere with soft contact lens wear.
* Prior corneal refractive surgery or corneal irregularity (e.g., keratoconus).
* Systemic disease, which might interfere with contact lens wear.
* Medication usage that may be associated with eye dryness.
* Use of any topical medication such as eye drops or ointment.
* Pregnant or lactating (by self-report).
* Aphakia.
* Grade 2 or greater of any of the following ocular surface signs: corneal edema, corneal vascularization, corneal staining, tarsal conjunctival changes or any other abnormality, which would normally contraindicate contact lens wear.
* Have participated in any other clinical trial or research in the two weeks prior to starting this study.

Ages: 15 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 157 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 157 subjects consented to participate in this study. Fifty-nine (59) subjects were determined to be ineligible. This allotted forty-nine (49) subjects randomly to each study arm for a total of 98 subjects enrolled.
Pre-assignment Details: Of the 59 identified as ineligible prior to group assignment, the majority were due to having a preexisting astigmatism.
Groups:
- Investigational Silicone Hydrogel Contact Lens: Subjects who were randomized to the study group wore contact lenses. These subjects were neophytes i.e., non-habitual contact lens wearers at the time of study enrollment.
- Spectacles: Subjects who randomized to this Control Group were non-habitual contact lens wearers and remained to be non-contact lens wearers.
Period: Baseline and Dispensed
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Started | 49 | 49
Completed | 47 | 49
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: 2-Week Visit
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Started | 47 | 49
Completed | 46 | 49
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: 1-Month Visit
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Started | 46 | 49
Completed | 44 | 49
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: 3-Month Visit
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Started | 44 | 49
Completed | 42 | 49
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Period: 6-Month Visit
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Started | 42 | 49
Completed | 34 | 40
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 6 | 7
Not completed — Lost to Follow-up | 2 | 2
Period: 1-Year Visit
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Started | 34 | 40
Completed | 29 | 37
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Population: Baseline participants were those who were randomly assigned to a study arm and started the study.
Groups:
- Investigational Silicone Hydrogel Contact Lens: Subjects randomized to the study arm wearing contact lenses. These subjects are considered neophytes and are non-habitual wearers. Test Group.
- Spectacles: Subjects are randomized to this Control Group.
- Total: Total of all reporting groups
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.57 (6.67) | 23.31 (6.08) | 22.94 (6.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 49
  Male | 21 | 28 | 49
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98

OUTCOME MEASURES:

1. Primary Outcome: Papillary Conjunctivitis
Description: Swelling of the papillary (Papillary conjunctivitis) area of the eye was assessed using a slit-lamp. Comparison between the two study arms will be assessed using data generated from a slit-lamp examination, using an Efron scale with 0.1 unit increments. The Efron scale has a range of 0 (normal) to 4 (Severe) and is subjectively assessed for 0.1 increments by the clinician, with the higher the magnitude of the number the worse the score.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the study groups, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Number analyzed (Participants) | 29 | 37
units on a scale | 0.98 [0.83 to 1.14] | 0.47 [0.32 to 0.61]

2. Primary Outcome: Conjunctival Hyperemia
Description: Comparison of the amount of redness in the conjunctival area of the eye, between the two study arms will be assessed using data generated from a slit-lamp examination, using an Efron scale with 0.1 unit increments. The Efron scale has a range of 0 (normal) to 4 (Severe) and is subjectively assessed for 0.1 increments by the clinician, with the higher the magnitude of the number the worse the score.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the study groups, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Number analyzed (Participants) | 29 | 37
units on a scale | 0.26 [0.13 to 0.39] | 0.28 [0.17 to 0.39]

3. Primary Outcome: Limbal Hyperemia
Description: Swelling of the vessels in the limbal area of the eye using a slit lamp. Comparison between the two study arms will be assessed using data generated from a slit-lamp examination, using an Efron scale with 0.1 unit increments. The Efron scale has a range of 0 (normal) to 4 (Severe) and is subjectively assessed for 0.1 increments by the clinician, with the higher the magnitude of the number the worse the score.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the study groups, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Number analyzed (Participants) | 29 | 37
units on a scale | 0.56 [0.45 to 0.67] | 0.30 [0.19 to 0.40]

4. Primary Outcome: Corneal Staining
Description: Abrasions in the cornea area of the eye using a slit lamp. Comparison between the two study arms will be assessed using data generated from a slit-lamp examination, using an Efron scale with 0.1 unit increments.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the study groups, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Efron Scale (0.1 Unit increments)
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Number analyzed (Participants) | 29 | 37
Efron Scale (0.1 Unit increments) | 0.26 [0.21 to 0.30] | 0.12 [0.07 to 0.16]

5. Primary Outcome: Conjunctival Staining
Description: Mild abrasions of the conjunctival area of the eye. Comparison between the two study arms will be assessed using data generated from a slit-lamp examination, using an Efron scale with 0.1 unit increments. The Efron scale has a range of 0 (normal) to 4 (Severe) and is subjectively assessed for 0.1 increments by the clinician, with the higher the magnitude of the number the worse the score.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the study groups, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Number analyzed (Participants) | 29 | 37
units on a scale | 1.41 [1.24 to 1.58] | 0.39 [0.24 to 0.55]

6. Primary Outcome: Corneal Neovascularization
Description: New vascularization of the Cornea. Comparison between the two study arms will be assessed using data generated from a slit-lamp examination, using an Efron scale with 0.1 unit increments. The Efron scale has a range of 0 (normal) to 4 (Severe) and is subjectively assessed for 0.1 increments by the clinician, with the higher the magnitude of the number the worse the score.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the study groups, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Number analyzed (Participants) | 29 | 37
units on a scale | 0.30 [0.25 to 0.34] | 0.09 [0.05 to 0.13]

7. Primary Outcome: Differences in Subjective Comfort From the Contact Lens User Experience (CLUE) Questionnaire
Description: The subjective comfort questionnaire CLUE, assesses the overall lens comfort. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response, with a range of 0-120. The differences between: (final visit and first visit) and then (final visit and 6 months) are reported.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the test group, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Investigational Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 29
units on a scale
  Comparison of First Visit - Last Visit | -4.97 [-12.26 to 2.32]
  Comparison of 6-Month Visit - Last Visit | 0.62 [-7.00 to 8.24]

8. Secondary Outcome: Comfortable Wearing Time
Description: Average numbers of overall average daily contact lens wear hours and average daily comfortable wear hours as reported at each follow-up visit.
Time Frame: 1 Year
Population: Subjects analyzed were those who were enrolled, randomized to the test group, and completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Investigational Silicone Hydrogel Contact Lens
Number analyzed (Participants) | 29
Hours | 10.25 [9.79 to 10.72]

ADVERSE EVENTS:
Arm/Group | Investigational Silicone Hydrogel Contact Lens | Spectacles
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication required agreement and written authorization from the Sponsor